CLINICAL TRIAL: NCT04837950
Title: Changes in Pleural Cavity Volume and Surgical Exposure Through Suture Retraction of the Diaphragm During VATS Procedures
Brief Title: Changes in Pleural Cavity Volume and Surgical Exposure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Peter B Licht, MD Professor, Odense University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 20/44867
Record Dates: First submitted 2020-11-09; First posted 2021-04-08 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Thoracic Cancer

STUDY DESIGN:
Intervention Model Description: During video-assisted thoracoscopic surgery a diaphragmatic traction-suture is placed posteriorly at the border between the central tendinous part and the peripheral muscular part. Body temperate saline solution is then poured into the pleural cavity until the cavity is filled up to the soft-tissue retractor in the utility port. The volume of saline in the pleural cavity is then measured and registered before and after distal contraction of the diaphragmatic traction suture through the camera port. Subsequently the surgeon will be asked to evaluate and rate the surgical field visual overview, before and after contraction of the suture. Furthermore, anonymized video recordings focusing on the pleural cavity visual overview before and after distal contraction of the suture, will be presented to specialist thoracic surgeons for a blinded evaluation.
Who Masked: Participant
Masking Description: Volume of saline in pleural cavity and surgical field overview before and after pulling traction suture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before pulling diaphragmatic suture (Experimental): Measurement of pleural cavity volume and visual overview before pulling diaphragmatic suture
  Interventions: Procedure: Diaphragmatic traction-suture
- After pulling diaphragmatic suture (Experimental): Measurement of pleural cavity volume and visual overview after pulling diaphragmatic suture
  Interventions: Procedure: Diaphragmatic traction-suture

INTERVENTIONS:
Procedure: Diaphragmatic traction-suture — Measurement of pleural cavity volume before pulling the diaphragmatic traction-suture Measurement of pleural cavity volume after pulling the diaphragmatic traction-suture

SUMMARY:
The investigators want to investigate if a diaphragmatic traction-suture affects the pleural cavity volume, as well as improves visual overview of a surgical field during minimally invasive thoracic surgery.

DETAILED DESCRIPTION:
A visually good surgical field is essential in performing safe and optimal dissection of anatomical structures during Video Assisted Thoracoscopic Surgery (VATS). A number of patients referred to VATS-surgery appear with an elevated diaphragm, reducing visibility and complicating safe surgical techniques, thus entailing conversion from VATS into an open Thoracotomy. Some surgeons handle the decreased visibility due to an elevated diaphragm by increasing the amount of ports during VATS. Others have benefited from attaching a traction suture on the diaphragmatic posterior tendinous part, thus flatting the diaphragmatic dome when the suture is tightly retracted through the camera-port. It turns out that most thoracic surgery clinics are not familiar with this technique. There are also no articles regarding this topic in medical literature. We want to investigate if the diaphragmatic traction-suture affects the pleural cavity volume, as well as improves visual overview of a surgical field during minimally invasive thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* known or suspected lung cancer
* scheduled for VATS-surgery
* perioperative finding of elevated diaphragma

Exclusion Criteria:

* not willing to give informed consent.
* perioperative finding of pleural adherences
* perioperative finding without an elevated diaphragma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Pleural cavity volume before | 1 minute after applying the traction suture
  Pleural cavity volume (ml) before distal retraction of the diaphragmatic traction suture.
Pleural cavity volume after | 2 minute after applying the traction suture
  Pleural cavity volume (ml) after distal retraction of the diaphragmatic traction suture.

SECONDARY OUTCOMES:
Visual overview | 1 minute after applying the traction suture
  The surgeon's evaluation of the surgical field visual overview before and after distal retraction of the diaphragmatic traction suture using a numeric rating scale (1-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Dept Cardiothorcic Surgery, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dittberner FA, Ladegaard L, Licht PB. A Diaphragmic Traction Suture Increases Pleural Cavity Volume and Surgical Field Overview During Video-Assisted Thoracoscopic Surgery. World J Surg. 2022 Jan;46(1):259-264. doi: 10.1007/s00268-021-06329-4. Epub 2021 Sep 29. PMID 34586461